CLINICAL TRIAL: NCT03745222
Title: A PHASE 3, RANDOMIZED, BLINDED, PLACEBO-CONTROLLED STUDY OF TISLELIZUMAB (BGB-A317) PLUS CHEMORADIOTHERAPY FOLLOWED BY TISLELIZUMAB MONOTHERAPY IN NEWLY DIAGNOSED, STAGE III SUBJECTS WITH LOCALLY ADVANCED, UNRESECTABLE NON-SMALL CELL LUNG CANCER
Brief Title: A Study of Tislelizumab (BGB-A317) Plus Chemoradiotherapy Followed by Tislelizumab Monotherapy in Newly Diagnosed, Stage III Subjects With Locally Advanced, Unresectable Non-small Cell Lung Cancer
Acronym: RATIONALE001
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: BeiGene and Celgene Corporation terminated the parties' global collaboration for the compound, pending the acquisition of Celgene by Bristol Myers Squibb
Sponsor: Celgene (Industry)
Collaborators: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BGB-A317-NSCL-001; U1111-1216-4294 (Other: WHO); 2018-001132-22 (EudraCT Number)
Record Dates: First submitted 2018-11-09; First posted 2018-11-19 (Actual); Results first posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Locally Advanced, Unresectable Non-Small Cell Lung Cancer; Non-Small Cell Lung Cancer; NSCLC; Randomized; BGB-A317; Tislelizumab; PD-1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; Chemoradiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1:Tislelizumab + cCRT followed by tislelizumab monotherapy (Experimental): Tislelizumab 200 mg is administered by intravenous (IV) administration and given together upfront with concurrent platinum-based chemoradiotherapy (cCRT) for the first 6 weeks, followed by tislelizumab 200 mg by IV adminstration monotherapy. The standard platinum-based chemotherapy options include carboplatin/ paclitaxel and cisplatin/etoposide
  Interventions: Drug: Tislelizumab; Drug: Concurrent chemoradiotherapy (cCRT)
- Arm 2: Placebo + cCRT followed by tislelizumab monotherapy (Experimental): Placebo is given with concurrent platinum-based chemoradiotherapy (cCRT) for the first 6 weeks, followed by tislelizumab 200 mg by IV administration monotherapy. The standard platinum-based chemotherapy options include carboplatin/paclitaxel and cisplatin/etoposide.
  Interventions: Drug: Tislelizumab; Drug: Concurrent chemoradiotherapy (cCRT); Other: Placebo
- Arm 3: Placebo + cCRT followed by placebo monotherapy (Placebo Comparator): Placebo is given with concurrent platinum-based chemoradiotherapy (cCRT) for the first 6 weeks, followed by placebo monotherapy. The standard platinum-based chemotherapy options include carboplatin/paclitaxel and cisplatin/etoposide.
  Interventions: Drug: Concurrent chemoradiotherapy (cCRT); Other: Placebo

INTERVENTIONS:
Drug: Tislelizumab — PD-1 inhibitor (monoclonal antibody against PD-1)
  Other Names: BGB-A317
  Arms: Arm 1:Tislelizumab + cCRT followed by tislelizumab monotherapy; Arm 2: Placebo + cCRT followed by tislelizumab monotherapy
Drug: Concurrent chemoradiotherapy (cCRT) — Chemotherapy options include carboplatin/paclitaxel and cisplatin/etoposide per standard of care. Radiotherapy will also be given concurrently with chemotherapy.
Other: Placebo — Placebo
  Arms: Arm 2: Placebo + cCRT followed by tislelizumab monotherapy; Arm 3: Placebo + cCRT followed by placebo monotherapy

SUMMARY:
This is a Phase 3, randomized, double-blind, placebo-controlled multicenter global study designed to compare the efficacy and safety of tislelizumab in combination with concurrent chemoradiotherapy (cCRT) followed by tislelizumab monotherapy versus cCRT alone, and tislelizumab given sequentially after cCRT versus cCRT alone, in newly diagnosed stage III subjects with locally advanced, unresectable non-small cell lung cancer (NSCLC). The primary endpoint is centrally-assessed progression free survival (PFS) in the intent-to-treat (ITT) population. .

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed, histologically confirmed, locally advanced, stage III unresectable non small cell lung cancer (NSCLC).

   Staging will be confirmed at screening by positron emission tomography-computed tomography (PET/CT) and brain imaging by magnetic resonance imaging (MRI) or computed tomography (CT) with contrast.
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
3. Epidermal growth factor receptor (EGFR) mutation and anaplastic lymphoma kinase (ALK) gene translocation status available prior to randomization.
4. Provision of fresh or archival tumor tissue or discussion with Sponsor.
5. Adequate hematologic and end-organ function.

Exclusion Criteria:

1. Prior therapies including those targeting PD-1 or PD-L1 or chemotherapy, radiation, targeted therapy, biologic therapy, immunotherapy or investigational agent used to control non-small cell lung cancer (NSCLC).
2. History of severe hypersensitivity reactions to other monoclonal antibodies or any contraindication to the planned chemotherapy regimen.
3. History of, or ongoing, interstitial lung disease; pneumonitis requiring steroids; or clinically significant pericardial effusion.
4. Any active malignancy less than or equal to 2 years before randomization, with the exception of non-small cell lung cancer (NSCLC) and any locally recurring cancer that has been treated curatively.
5. Severe chronic or active infections including those requiring systemic antibacterial, antifungal or antiviral therapy; known human immunodeficiency virus (HIV) infection; untreated chronic hepatitis B or chronic hepatitis B virus carries or active hepatitis C; or active autoimmune disease.
6. Prior allogeneic stem cell transplantation or organ transplantation.
7. Significant cardiovascular disease or other condition which places the patient at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Nguyen, MD, Study Director — Celgene
Locations (164):
- United States (14):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Cancer Specialists of North Florida - Jacksonville, Jacksonville, Florida
  - Bond Clinic, P.A., Winter Haven, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Appalachian Regional Healthcare, Inc., Hazard, Kentucky
  - Norton Healthcare - Norton Cancer Institute, Louisville, Kentucky
  - Center For Cancer and Blood Disorders, Bethesda, Maryland
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Dayton Physicians, LLC, Kettering, Ohio
  - Mercy Health Youngstown Hospital, LLC, Youngstown, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Millennium Oncology, Houston, Texas
  - Medical Oncology Associates, P.S., Spokane, Washington
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
- Jewish General Hospital, Montreal, Quebec, Canada
- China (33):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Chinese PLA General Hospital / 307 Hospital, Beijing
  - Beijing Cancer Hospital - Beijing Institute for Cancer Research, Beijing
  - Bengbu Medical College - First Affiliated Hospital, Bengbu Shi
  - Jilin Province Cancer Hospital, Changchun
  - First Hospital of Jilin University, Changchun
  - Central South University - Xiangya School of Medicine - Hunan Cancer Hospital, Changsha
  - Central South University - Xiangya School of Medicine - Hunan Cancer Hospital, Changsha-shi
  - Sichuan Cancer Hospital & Institute, Chengdu
  - Sichuan University - West China Hospital, Chengdu
  - Foshan First People's Hospital, Foshan
  - Cancer Center of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Zhejiang University School of Medicine - The Second Affiliated Hospital, Hangzhou
  - Zhejiang Medical University - Zhejiang Cancer Hospital, Hangzhou
  - The First Affiliated Hospital of Harbin Medical University, Harbin
  - Yunnan Cancer Hospital, Kunming
  - Guangxi Tumour Institute and Hospital, Nanning
  - Nantong Tumor Hospital, Nantong
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai Chest Hospital, Shanghai Shi
  - Chongqing Cancer Hospital, Shapingbaqu
  - Liaoning Cancer Hospital & Institute, Shenyang
  - The First Hospital of Xinjiang Medical University, Ürümqi
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Zhongnan Hospital of Wuhan University, Wuhan
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - First Hospital of Xiamen, Xiamen
  - Fujian Medical University - Fujian Provincial Cancer Hospital, Xidajie
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Zhengzhou University (ZZU) - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Finland (2):
  - Tampereen yliopistollinen sairaala, Tampere
  - Turku University Hospital, Turku
- France (3):
  - Centre Francois Baclesse, Caen
  - Clinique Victor Hugo, Le Mans
  - Institut de Cancerologie de l'Ouest (ICO) - Saint-Herblain, Saint-Herblain
- Germany (13):
  - Medical Study Company NORD-WEST GmbH Oncology Aurich, Aurich
  - Helios Klinikum Emil Von Behring, Berlin
  - Kliniken der Stadt Koln gGmbH - Krankenhaus Merheim, Cologne
  - Florence Nightingale KH der Kaiserwerther Diakonie, Düsseldorf
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Asklepios Fachkliniken Muenchen Gauting, Gauting
  - Oncological practice Goslar, Goslar
  - Evangelisches Krankenhaus Hamm, Hamm
  - Health Nordhessen Holding AG - Klinikum Kassel - Medical Clinic IV, Kassel
  - Klinik Loewenstein gGmbH, Löwenstein
  - LMU Klinikum der Universität, München
  - St. Antonius-Hospital, Schweiler
  - Medizinische Studiengesellschaft Nord-West, Westerstede
- Greece (10):
  - Sotiria Chest Hospital of Athens, Athens
  - IASO General, Athens
  - University General Hospital of Heraklion, Heraklion
  - Agioi Anargyroi Cancer Hospital, Kifissia
  - Metaxa Cancer Hospital of Piraeus, Piraeus
  - Interbalkan Medical Center of Thessaloniki, Pylaia
  - University General Hospital of Patras, Rio Patras
  - Bioclinic Thessaloniki Galinos clinic, Thessaloniki
  - EUROMEDICA General Clinic of Thessaloniki, Thessaloniki
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
- Hungary (2):
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
  - Pulmonary Institute Torokbalint, Törökbálint
- Ireland (3):
  - Beacon Hospital, Dublin
  - St James Hospital, Dublin
  - MidWestern Regional Hospital, Limerick
- Italy (5):
  - Azienda Ospedaliero - Universitaria Policlinico - Vittorio Emanuele - Ospedale Gaspare Rodolico, Catania
  - IRCCS AziendaOspedaliera Universitaria San Martino, Genova
  - Istituto Scientifico Romagnolo Per Lo Studio e La Cura Dei Tumori (I.R.S.T.), Meldola
  - Universita Campus Bio-Medico di Roma, Roma
  - Istituto Nazionale Tumori Regina Elena di Roma, Roma
- Japan (16):
  - Osaka Prefectural Medical Center for Respiratory and Allergic Diseases, Habikino-shi
  - Kansai Medical University Hospital, Hirakata-shi
  - Hiroshima University Hospital, Hiroshima
  - Kanazawa University Hospital, Kanazawa
  - Matsusaka Municipal Hospital, Matsusaka-shi
  - Toranomon Hospital, Minatoku
  - Iwate Medical University Hospital, Morioka
  - National Hospital Organization - Nagoya Medical Center, Nagoya
  - Nagoya University Hospital, Nagoya
  - Niigata Cancer Center Hospital, Niigata
  - Osaka City University Hospital, Osaka
  - Gunma Prefectural Cancer Center, Ōta-ku
  - Kitasato University Hospital, Sagamihara
  - Sendai Kousei Hospital, Sendai
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama
  - Yokohama Municipal Citizen's Hospital, Yokohama
- Netherlands (2):
  - Vrije Universiteit Medisch Centrum (VUMC), Amsterdam
  - Gelre Hospitals, Zutphen
- New Zealand (2):
  - Waikato Hospital, Hamilton
  - Tauranga Hospital, Tauranga
- Poland (4):
  - Centrum Onkologii im. prof. Franciszka Lukaszczyka w Bydgoszczy, Bydgoszcz
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej-Curie, Gliwice
  - Med Polonia Sp. z o.o. NSZOZ, Poznan
  - Centrum Onkologii-Instytut im.Marii Sklodowskiej-Curie, Warsaw
- Portugal (7):
  - Hospital Prof. Doutor Fernando Fonseca, Amadora
  - Centro Hospitalar E Universitario de Coimbra EPE, Coimbra
  - Centro Hospitalar do Alto Ave, Hospital da Senhora da Oliveira Guimaraes, Guimarães
  - CUF Descobertas Hospital, Lisbon
  - Centro Hospitalar do Porto - Hospital de Santo António, Porto
  - CUF Porto Hospital, Porto
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil Epe, Porto
- Romania (7):
  - Oncology Institute Professor Doctor Alexandru Trestioreanu, Bucharest
  - Prof. Dr. I. Chiricuta Institute of Oncology, Cluj-Napoca
  - Medisprof SRL, Cluj-Napoca
  - Sf. Apostol Andrei Constanta Emergency Clinical County Hospital, Constanța
  - Oncology Center Sfantul Nectarie, Craiova
  - Life Search SRL, Timișoara
  - Oncocenter Clinical Oncology, Timișoara
- Russia (7):
  - Principal Military Clinical Hospital n.a. N.N. Burdenko, Moscow
  - Omsk Regional Oncology Center, Omsk
  - Ryazan State Medical University n.a. I.P. Pavlov, Ryazan
  - Clinical Hospital of the Russian Academy of Sciences, Saint Petersburg
  - GBUZ Saint Petersburg Clinical Research Center of Specialized Types of Care (Oncology), Saint Petersburg
  - Research Oncology Institute of Rosmed Technologies n.a. prof. N.N. Petrov, Saint Petersburg
  - Mordovia State University, Saransk
- Singapore (2):
  - National University Hospital, Singapore
  - Raffles Hospital, Singapore
- South Korea (4):
  - Chungbuk National University Hospital, Cheongju-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Ajou University Hospital, Suwon
- Spain (10):
  - Hospital Universitario a Coruna, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Germans Trias i Pujol, Barcelona
  - Insular-Maternal and Child University Hospital Complex, Las Palmas de Gran Canaria
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro-Majadahonda, Majadahonda, Madrid
  - Hospital General Carlos Haya, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Taiwan (5):
  - Buddhist Dalin Tzu Chi General Hospital, Dalin
  - E-DA Hospital, Kaohsiung City
  - Kaohsiung Medical University Hospital, Kaohsiung, San Ming Dist.
  - Chang Gung Medical Foundation, Kaohsiung Memorial Hospital, Niao-Sung Hsiang Kaohsiung County
  - National Taiwan University Hospital, Taipei, Zhongzheng Dist.
- United Kingdom (10):
  - University Hospitals Birmingham NHS Foundation Trust - Queen Elizabeth Hospital, Birmingham
  - East Suffolk and North Essex NHS Foundation Trust - Colchester Hospital, Colchester
  - University College London Hospitals NHS Foundation Trust - University College Hospital, London
  - Guys Hospital, London
  - Royal Marsden Hospital, London
  - Maidstone and Tunbridge Wells NHS Trust - Maidstone Hospital, Maidstone
  - Manchester University NHS Foundation Trust - Wythenshawe Hospital - North West Lung Centre, Manchester
  - The Hillingdon Hospitals NHS Foundation Trust - Mount Vernon Hospital, Northwood
  - Sheffield Teaching Hospitals NHS Foundation Trust - Weston Park Hospital, Sheffield South Yorkshire
  - Royal Cornwall Hospitals Trust, Truro

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant was enrolled in the United States before the study was terminated.
Groups:
- Tislelizumab + Concurrent Chemoradiotherapy -Tislelizumab: Participants were to receive 2 cycles of tislelizumab 200 mg by intravenous (IV) infusion every 3 weeks (Q3W) with concurrent chemoradiotherapy (cCRT), followed by monotherapy with tislelizumab 200 mg IV Q3W until disease progression, death, unacceptable toxicity, subject or physician decision, withdrawal of consent or treatment discontinuation for another reason.
- Placebo + Concurrent Chemoradiotherapy -Tislelizumab: Participants were to receive 2 cycles of identically matching placebo by IV infusion Q 3 weeks with cCRT, followed by monotherapy with tislelizumab 200 mg IV Q 3W until disease progression, death, unacceptable toxicity, subject or physician decision, withdrawal of consent or treatment discontinuation for another reason.
- Placebo + Concurrent Chemoradiotherapy - Placebo: Participants were to receive 2 cycles of identically matching placebo by IV infusion Q 3 weeks with cCRT, followed by monotherapy with placebo IV Q 3W until disease progression, death, unacceptable toxicity, subject or physician decision, withdrawal of consent or treatment discontinuation for another reason.
Period: Overall Study
Arm/Group | Tislelizumab + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy - Placebo
Started | 0 | 1 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat Population included all randomized participants regardless of whether the participant received any study drug or had any efficacy assessments performed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tislelizumab + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy - Placebo | Total
Number analyzed (Participants) | 0 | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 |  | 0
  Between 18 and 65 years |  | 1 |  | 1
  >=65 years |  | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival was defined as the time from the date of randomization to the date of the first objectively tumor progression as assessed by the blinded independent central review per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 criteria (documented by radiological assessment) or death (any cause) on or prior to the clinical cut-off date, which ever occurred first. Stable disease-neither sufficient shrinkage to qualify for PR nor sufficient increase of lesions to qualify for Progressive disease (PD)• Progressive Disease- At least a 20% increase in the sum of diameters of target lesions from nadir.
Time Frame: Up to approximately 5 years; date of randomization to the date of tumor progression or death; until study withdrawal date of 26 June 2019
Population: The study was terminated. The number of participants and the data collection period were not sufficient for statistical analysis. The patient withdrew consent.
Arm/Group | Tislelizumab + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy - Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time between randomization of treatment and death from any cause.
Time Frame: Up to approximately 5 years; date of randomization to date of death from any cause.
Population: as for outcome 1
Arm/Group | Tislelizumab + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy - Placebo
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Overall Survival at 24 Months
Description: Overall survival was defined as the time between randomization of treatment and death from any cause.
Time Frame: Up to approximately 24 months
Population: as for outcome 1
Arm/Group | Tislelizumab + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy - Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Percentage of Participants Who Achieved a Best Overall Response of Complete Response or Partial Response
Description: Overall Response was defined as percentage of participants who had a radiologic confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) guidelines, between Day 1 of treatment and subsequent anti-cancer therapy, death or study discontinuation. Complete response was defined as the disappearance of all target lesions; partial response (PR) is defined as at least a 30% decrease in the sum of diameters of target lesions from baseline; stable disease-neither sufficient shrinkage to qualify for PR nor sufficient increase of lesions to qualify for progressive disease (PD).
Time Frame: Up to approximately 5 years
Population: as for outcome 1
Arm/Group | Tislelizumab + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy - Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Duration of Response
Description: Duration of Response is defined as the time from the first occurrence of a documented objective response to the time of relapse, as determined by blinded independent central review per RECIST v1.1, or death from any cause, whichever comes first.
Time Frame: Up to approximately 5 years
Population: as for outcome 1
Arm/Group | Tislelizumab + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy - Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants Alive and Progression-Free at 12 Months (APF12)
Description: Progression-free survival was defined as the time from the date of randomization to the date of the first objectively tumor progression as assessed by the blinded independent central review per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 criteria (documented by radiological assessment) or death (any cause) on or prior to the clinical cut-off date, which ever occurred first
Time Frame: Up to 12 months
Population: as for outcome 1
Arm/Group | Tislelizumab + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy - Placebo
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants Alive and Progression-free at 18 Months (APF18)
Description: as for outcome 6
Time Frame: Up to approximately 18 months
Population: as for outcome 1
Arm/Group | Tislelizumab + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy - Placebo
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Time to Distant Metastasis (TTDM)
Description: TTDM was defined as the time from the date of randomization until the first date of distant metastasis or death in the absence of distant metastasis. Distant metastasis was defined as any new lesion that is outside of the radiation field according to RECIST v1.1 or proven by biopsy.
Time Frame: Up to approximately 5 years
Population: as for outcome 1
Arm/Group | Tislelizumab + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy - Placebo
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs include any adverse events (AEs) that had an onset date or a worsening in severity from baseline on or after the first dose of study drug up to 30 days following study drug discontinuation or initiation of new anticancer therapy, whichever occurred first. TEAEs also included all immune-related AEs recorded up to 90 days after the last dose of tislelizumab or placebo, regardless of whether or not the particpant started a new anticancer therapy. In addition, any serious AE with an onset date more than 30 days after the last dose of study drug that is assessed by the investigator as related to study drug were considered a TEAE."
Time Frame: From first dose of study drug up to study withdrawal date of 26 June 2019; 15 days.
Population: Safety population includes participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Tislelizumab + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy - Placebo
Number analyzed (Participants) | 0 | 1 | 0
Participants
  ≥ 1 TEAE |  | 1 |
  ≥ 1 Treatment Related TEAE |  | 1 |

10. Secondary Outcome: Number of Participants With Lung Cancer Symptoms Assessed by the Corresponding Domains of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC-QLQ-C30) and Lung-Cancer Specific QLQ-LC13
Description: The EORTC QLQ-C30 is a 30-item, questionnaire assessing quality of life (QoL), psychosocial burden and physical symptoms. It is classified into 15 domains: 5 functional subscales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning); 3 multi-item symptom subscales (fatigue, nausea/vomiting, and pain); each item is measured on a 4 point response scale; (not at all, a little, quite a bit, very much), with the exception of the 2 items measuring global health and QoL, (measured on a 7-point response scale). Scores are linearly transformed to 0 to 100 scores. Scores vary from 0 (worst) to 100 (best) for the functional dimensions and GHS, and from 0 (best) to 100 (worst) for the symptom dimensions; higher scores = better QoL, better functioning, or more severe symptoms, respectively. The LC13 covers 13 typical symptoms of lung cancer patients, such as coughing, pain, dyspnea, sore mouth, peripheral neuropathy, and hair loss.
Time Frame: Up to approximately 5 years
Population: as for outcome 1
Arm/Group | Tislelizumab + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy - Placebo
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants Who Would Have Continued on to Monotherapy Phase
Description: Included the percentage of participants who would have received at least one dose of tislelizumab or placebo in the monotherapy phase before progression.
Time Frame: Up to approximately 5 years
Population: as for outcome 1
Arm/Group | Tislelizumab + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy - Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to study withdrawal date of 26 June 2019; 15 days.
Description: No serious adverse events or deaths occurred during the course of the study,
Arm/Group | Tislelizumab + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy -Tislelizumab | Placebo + Concurrent Chemoradiotherapy - Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tislelizumab + Concurrent Chemoradiotherapy -Tislelizumab (N=0) | Placebo + Concurrent Chemoradiotherapy -Tislelizumab (N=1) | Placebo + Concurrent Chemoradiotherapy - Placebo (N=0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
MUSCLE CRAMPING (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission and defer publication to permit patent applications.

DOCUMENTS (2):
  • Study Protocol (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT03745222/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT03745222/SAP_001.pdf